CLINICAL TRIAL: NCT01012947
Title: Cognitive Health Promotion Project in the Community
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Chang Hyung Hong, Associate Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AjouU
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-01

CONDITIONS: Alteration of Cognitive Function; Dietary Modification
Keywords: MMSE; activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Lifestyle Counseling Usual Care (Experimental): Usual care participants in the group A received no additional services.
  Interventions: Behavioral: Lifestyle Counseling Usual Care
- Lifestyle Counseling Telephone, Bimonth (Experimental): Participants in the group B received bimonthly telephonic care management based on manual.
  Interventions: Behavioral: Lifestyle Counseling Telephone, Bimonth
- Lifestyle Counseling Telephone, Month (Experimental): Participants in the group C received monthly the same telephonic care management and educational materials as those in the group B.
  Interventions: Behavioral: Lifestyle Counseling Telephone, Month
- Lifestyle Counseling Visit, Bimonth (Experimental): Participants in the group D received health educator-initiated visit counseling bimonthly.
  Interventions: Behavioral: Lifestyle Counseling Visit, Bimonth
- Lifestyle Counseling Visit, Reward (Experimental): Participants in the group E received health educator-initiated visit counseling bimonthly and reward.
  Interventions: Behavioral: Lifestyle Counseling Visit, Reward

INTERVENTIONS:
Behavioral: Lifestyle Counseling Usual Care — Usual care participants in the group A received no additional services.
  Other Names: Group A usual care
  Arms: Lifestyle Counseling Usual Care
Behavioral: Lifestyle Counseling Telephone, Bimonth — Participants in the group B received bimonthly telephonic care management based on manual.
  Other Names: Group B bimonthly telephone
  Arms: Lifestyle Counseling Telephone, Bimonth
Behavioral: Lifestyle Counseling Telephone, Month — Participants in the group C received monthly the same telephonic care management and educational materials as those in the group B.
  Other Names: Group C monthly telephone
  Arms: Lifestyle Counseling Telephone, Month
Behavioral: Lifestyle Counseling Visit, Bimonth — Participants in the group D received health educator-initiated visit counseling bimonthly.
  Other Names: Group D bimonthly visit
  Arms: Lifestyle Counseling Visit, Bimonth
Behavioral: Lifestyle Counseling Visit, Reward — Participants in the group E received health educator-initiated visit counseling bimonthly and reward.
  Other Names: Group E bimonthly visit and reward
  Arms: Lifestyle Counseling Visit, Reward

SUMMARY:
This study was based on baseline data derived from a large prospective study called the Suwon Project (SP), a cohort comprising random clustering samples of elderly people, all of whom are ethnic Koreans aged over 60 years.

DETAILED DESCRIPTION:
There is growing evidence supporting the protective effect of health behaviors against cognitive decline and dementia in older persons. With this increasing evidence and a better understanding of the underlying mechanisms, lifestyle modification is likely to be increasingly promoted as a convincing strategy for maintaining cognitive health in later life.

The study protocol included cognitive screening through the Korean version of the Mini-Mental State Examination (K-MMSE), which has been validated for the Korean-speaking population ({YW, 1997 #88}Kang YW et al., 1997), recording of the subject's medical history. A Korean study in the community defined the cut-off point of K-MMSE score during the screening of dementia as 17/18 points; the sensitivity and specificity of the findings were 91% and 86%, respectively ({YW, 1997 #88}Kim et al., 2003). Based on these results, we defined cognitive impairment (CI) as the group that had a K-MMSE score lower than 17, and not cognitive impairment (NCI) was defined as the group that had a K-MMSE score higher than 18.

ELIGIBILITY:
Inclusion Criteria:

* more than 60 years old

Exclusion Criteria:

* those with a history of significant hearing or visual impairment that rendered participation in the interview difficult
* those with a history of neurological disorders (e.g., stroke, Parkinson's disease, or active epilepsy)
* those with psychiatric illness (e.g., schizophrenia, mental retardation, severe depression, or mania)
* those taking psychotropic medications, or those with significant alcohol and other substance abuse.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1115 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chang Hyung Hong, MD PhD, Principal Investigator — Ajou University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted from August 2008 to December 2010 at a geriatric mental health community center in Suwon, south Korea. The center, which has been established since 2008 and has outreach sites throughout the districts, provides a range of social, health, educational, and recreational services for users of elderly groups.
Pre-assignment Details: Criteria for exclusion included severe visual or hearing impairment and a previous diagnosis of idiopathic Parkinson's disease, liver disease, alcoholism, or known terminal illness. Prior to initiating the study, we obtained a list of all senior citizen centers. A random number table was used to classify the intervention group.
Groups:
- Lifestyle Counseling A,Usual Care: Usual care participants received no additional services.
- Lifestyle Counseling B, Telephone, Bimonthly: Participants in the group B received bimonthly telephonic care management based on manual. Manager received training on a brief advice process, consisting of assessing activity level using a simple self-assessment tool; providing advice to increase activity and select a long-term goal.
- Lifestyle Counseling C, Telephone, Monthly: Participants in the group C received monthly the same telephonic care management and educational materials as those in the group B.
- Lifestyle Counseling D, Visit, Bimonthly: Participants in the group D received health educator-initiated visit counseling bimonthly.
- Lifestyle Counseling E, Visit, Reward: Participants in the group E received health educator-initiated visit counseling bimonthly. Participants in the group E received reward.
Period: Overall Study
Arm/Group | Lifestyle Counseling A,Usual Care | Lifestyle Counseling B, Telephone, Bimonthly | Lifestyle Counseling C, Telephone, Monthly | Lifestyle Counseling D, Visit, Bimonthly | Lifestyle Counseling E, Visit, Reward
Started | 212 | 215 | 241 | 211 | 236
Completed | 81 | 80 | 111 | 93 | 94
Not Completed | 131 | 135 | 130 | 118 | 142
Not completed — Lost to Follow-up | 131 | 135 | 130 | 118 | 142

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Counseling A,Usual Care | Lifestyle Counseling B, Telephone, Bimonthly | Lifestyle Counseling C, Telephone, Monthly | Lifestyle Counseling D, Visit, Bimonthly | Lifestyle Counseling E, Visit, Reward | Total
Number analyzed (Participants) | 212 | 215 | 241 | 211 | 236 | 1115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 212 | 215 | 241 | 211 | 236 | 1115
Age Continuous [Mean (Standard Deviation); unit: years] | 77.5 (1.9) | 76.5 (2.9) | 77.3 (1.7) | 77.9 (3.7) | 76.7 (2.1) | 77.1 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 174 | 188 | 170 | 172 | 861
  Male | 55 | 41 | 53 | 41 | 64 | 254
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 212 | 215 | 241 | 211 | 236 | 1115

OUTCOME MEASURES:

1. Primary Outcome: Change of Cognitive Function Measured by a Mini Mental State Examination Scores on a Scale According to Study Group
Description: The mini-mental state examination (MMSE) or Folstein test is a brief 30-point questionnaire test that is used to screen for cognitive impairment. It ranges from 0 to 30 points. The higher scores mean better outcome. It is also used to estimate the severity of cognitive impairment at a given point in time and to follow the course of cognitive changes in an individual over time, thus making it an effective way to document an individual's response to treatment.
  In the time span of about 10 minutes it samples various functions including arithmetic, memory and orientation.
Time Frame: baseline and 18 months
Population: The location of the survey was Suwon City, with a population of 1 million, located adjacent to Seoul, the nation's capital. The center, which has been established since 2008 and has outreach sites throughout the districts, provides a range of social, health, educational, and recreational services for users of elderly groups.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Counseling A,Usual Care | Lifestyle Counseling B, Telephone, Bimonthly | Lifestyle Counseling C, Telephone, Monthly | Lifestyle Counseling D, Visit, Bimonthly | Lifestyle Counseling E, Visit, Reward
Number analyzed (Participants) | 212 | 215 | 241 | 211 | 236
units on a scale | 23.3 (2.3) [21 to 28.8] | 23.8 (2.1) | 23.1 (1.0) | 23.7 (1.4) | 24.2 (0.7)

ADVERSE EVENTS:
Arm/Group | Lifestyle Counseling A,Usual Care | Lifestyle Counseling B, Telephone, Bimonthly | Lifestyle Counseling C, Telephone, Monthly | Lifestyle Counseling D, Visit, Bimonthly | Lifestyle Counseling E, Visit, Reward
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/215 | 0/241 | 0/211 | 0/236
Other Adverse Events (participants affected / at risk) | 0/212 | 0/215 | 0/241 | 0/211 | 0/236

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No